CLINICAL TRIAL: NCT00515216
Title: Pharmacogenomically Selected Treatment for Gastric and Gastroesophageal (GEJ) Tumors: A Phase II Study
Brief Title: Pharmacogenomically Selected Treatment for Gastric and Gastroesophageal Junction (GEJ) Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of Alabama at Birmingham (Other); University of North Carolina (Other); Washington University School of Medicine (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Craig Lockhart, Associate Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070433; R21CA123881 (NIH)
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
Keywords: Phase II; Gastric cancer; Gastroesophageal cancer; Metastatic; FOLFOX; Thymidylate synthase; Pharmacogenomic
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis | interventions — Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin/Leucovorin/5-FU (Experimental): "Good risk" patients with the TSER*2/*2 or *2/*3 genotype or low TS expression genotype received treatment of oxaliplatin, leucovorin given over 2 hours along with 5-FU given as intravenous push followed by 5-FU given as intravenous infusion of 46 hours. This treatment was repeated every 2 weeks.
  Interventions: Drug: 5-fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: 5-fluorouracil
  Other Names: 5-FU; Fluorouracil
Drug: Oxaliplatin
  Other Names: Eloxatin
Drug: Leucovorin
  Other Names: Wellcovorin; citrovorum factor; folinic acid; 5-formyl tetrahydrofolate

SUMMARY:
This study is for patients who have stomach cancer or cancer of the lower part of the esophagus that has spread to other organs. There are many different chemotherapy treatments for this type of cancer. At the present time, there is no general agreement on the way to choose the most beneficial therapy for an individual patient. Patients with different genetic backgrounds may respond differently to the same chemotherapy treatments. In this study the investigators will use a certain genetic difference in an important gene (thymidylate synthase or TS gene) to see whether treating patients who have a particular type of that gene will respond better to a standard chemotherapy regimen. The investigators are hoping that by treating patients according to their genes, that they may respond to treatment of their cancer better and it will help the investigators choose cancer treatments better in the future.

DETAILED DESCRIPTION:
Gastric and gastroesophageal junction (GEJ) cancers are a leading cause of cancer mortality. Despite the development of newer chemotherapies, the response rates and median survival in patients with these tumors has remained essentially stagnant. Defining host and molecular/biologic tumor characteristics to customize treatment may lead to improved survival outcomes. Retrospective studies have identified genetic markers that predict treatment outcome. However, there have been no prospective studies in gastric and GEJ cancer evaluating the clinical utility of these genetic factors. We hypothesize that genomically based treatment will improve the expected response rate in patients with gastric and GEJ cancers. We propose a prospective, multi-institutional Phase II clinical trial testing a germline polymorphism in the thymidylate synthase (TS) gene, the number of tandem repeats in the TS enhancer region (TSER) as a treatment selection marker. The polymorphic variant conferring three tandem repeats (TSER*3) has been associated with 5-FU resistance due to high tumor TS expression in comparison to the TSER*2 variant (two tandem repeats). The TSER*3 polymorphism is common (allelic frequency of 0.5-0.8). In the proposed study, we will prospectively genotype patients with gastric and GEJ cancers. Patients who are expected to be 5-FU sensitive (carrying a TSER*2 allele) will receive a 5-FU containing regimen (5-FU, leucovorin, oxaliplatin). Patients who are expected to be 5-FU resistant (homozygous for TSER*3) will not be included in the study. In completing this study, we will determine whether treatment selection based on germline TSER polymorphism status improves the response rate in patients with metastatic gastric and GEJ tumors. Additional correlative studies are proposed to identify confounding factors that may alter the expected outcomes of this treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction.
* Patients must have measurable disease.
* No prior therapy for metastatic disease. Prior neo-adjuvant or adjuvant therapy is permitted if the disease free interval has been longer than 6 months.
* Age ≥18 years.
* Life expectancy of greater than 3 months.
* ECOG (Eastern Cooperative Oncology Group) performance status greater than 2 (Karnofsky greater than 60%).
* Patients must have normal organ and marrow function.
* Not pregnant. Not breast feeding.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other chemotherapy agents.
* Patients with known active brain metastases. Patients with treated brain metastases are permitted if stable off steroids for at least 30 days.
* History of allergic reactions to 5-FU or oxaliplatin.
* Uncontrolled intercurrent illness.
* Patients with immune deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert C. Lockhart, M.D., Principal Investigator — Washington University School of Medicine; Laura Goff, M.D., Principal Investigator — Vanderbilt University Medical Center; Richard Goldberg, M.D., Principal Investigator — University of North Carolina; James Posey, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Washington University School of Medicine, St Louis, Missouri
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Goff LW, Thakkar N, Du L, Chan E, Tan BR, Cardin DB, McLeod HL, Berlin JD, Zehnbauer B, Fournier C, Picus J, Wang-Gillam A, Lee W, Lockhart AC. Thymidylate synthase genotype-directed chemotherapy for patients with gastric and gastroesophageal junction cancers. PLoS One. 2014 Sep 18;9(9):e107424. doi: 10.1371/journal.pone.0107424. eCollection 2014. PMID 25232828
- See also: Vanderbilt-Ingram Cancer Center — http://www.vicc.org
- See also: Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu
- See also: UNC Lineberger Comprehensive Cancer Center — http://cancer.med.unc.edu
- See also: University of Alabama at Birmingham . Comprehensive Cancer Center — http://www3.ccc.uab.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to participant enrollment in June 2008 and closed to participant enrollment in October 2010.
Groups:
- Oxaliplatin/Leucovorin/5-FU: "Good risk" patients with the TSER*2/*2 or *2/*3 genotype or low TS expression genotype
  Chemotherapy: 5-FU, leucovorin and oxaliplatin (FOLFOX)
Period: Overall Study
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Started | 26
Completed | 25
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 56 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 26
TSER genotypes [Number; unit: participants]
  TSER*2/*2 | 5
  TSER*2/*3 | 21
ECOG Performance Status [Number; unit: participants] — 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  participants
    0 | 5
    1 | 13
    2 | 8
Primary tumor type [Number; unit: participants]
  Gastric | 19
  Gastroesophageal junction | 7
Incidence of prior neoadjuvant or adjuvant therapy (>6 months) [Number; unit: percentage of participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: * ORR = complete response + partial response
  * Complete response - disappearance of all target and non-target lesions
  * Partial response - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 25
percentage of participants | 39.1 [22.2 to 59.2]

2. Secondary Outcome: Overall Survival
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 25
months | 11.4 [6.3 to 16.3]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progressive disease - at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 25
months | 6.2 [5.2 to 8.6]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR - complete response, partial response, and stable disease
  * Complete response - disappearance of all target and non-target lesions
  * Partial response - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
  * Stable disease - neither sufficient shrinkage to qualify for partial response not sufficient increase to qualify for progressive disease
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 25
percentage of participants | 95.7 [79.0 to 99.2]

5. Secondary Outcome: Tumor Specific Changes That May Alter Treatment Outcomes
Time Frame: 4 years
Population: This was not completed as the archived tumor samples were not of sufficient quality for DNA extraction or analysis.
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 0

6. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Partial Response)
Description: This outcome looks at what genotypes of the TYMS 5'-UTR TSER + G>C (rs34743033) gene had a partial tumor response.
Time Frame: 4 years
Population: 9 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 9
participants
  TYMS, TSER*2/*2 | 5
  TYMS, TSER*2/*3 (G) | 2
  TYMS, TSER*2/*3 (C) | 2

7. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Partial Response)
Description: This outcome looks at what genotypes of the TYMS 3'-UTR 1494delTTAAAG(6 bp) (rs34489327) gene had a partial tumor response.
Time Frame: 4 years
Population: 9 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 9
participants
  +6 bp/+6 bp | 5
  +6 bp/-6 bp | 4

8. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Partial Response)
Description: This outcome looks at what genotypes of the ERCC1 c.354C>T (rs11615) gene had a partial tumor response.
Time Frame: 4 years
Population: 9 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 9
participants
  C/C | 2
  C/T | 4
  T/T | 3

9. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Partial Response)
Description: This outcome looks at what genotypes of the ERCC2 c.2251A>C (rs13181) gene had a partial response.
Time Frame: 4 years
Population: 9 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 9
participants
  A/A | 5
  A/C | 3
  C/C | 1

10. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Partial Response)
Description: This outcome looks at what genotypes of the GSTP1 c.313A>G (rs1695) gene had a partial response.
Time Frame: 4 years
Population: 9 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 9
participants
  A/A | 4
  A/G | 3
  G/G | 2

11. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Partial Response)
Description: This outcome looks at what genotypes of the XRCC1 c.1196G>A (rs25487) gene had a partial response.
Time Frame: 4 years
Population: 9 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 9
participants
  A/A | 1
  G/A | 6
  G/G | 2

12. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Partial Response)
Description: This outcome looks at what genotypes of the MDR1 c.3435C>T (rs1045642) gene had a partial response.
Time Frame: 4 years
Population: 9 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 9
participants
  C/C | 0
  C/T | 9
  T/T | 0

13. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Stable Disease)
Description: This outcome looks at what genotypes of the TYMS 5'-UTR TSER + G>C (rs34743033) gene had stable disease.
Time Frame: 4 years
Population: 11 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 11
participants
  TYMS, TSER*2/*2 | 1
  TYMS, TSER*2/*3 (G) | 4
  TYMS, TSER*2/*3 (C) | 6

14. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Stable Disease)
Description: This outcome looks at what genotypes of the TYMS 3'-UTR 1494delTTAAAG(6 bp) (rs34489327) gene had stable disease.
Time Frame: 4 years
Population: 11 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 11
participants
  +6 bp/+6 bp | 6
  +6 bp/-6 bp | 5

15. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Stable Disease)
Description: This outcome looks at what genotypes of the ERCC1 c.354C>T (rs11615) gene had stable disease.
Time Frame: 4 years
Population: 11 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 11
participants
  C/C | 1
  C/T | 8
  T/T | 2

16. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Stable Disease)
Description: This outcome looks at what genotypes of the ERCC2 c.2251A>C (rs13181) gene had stable disease.
Time Frame: 4 years
Population: 11 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 11
participants
  A/A | 3
  A/C | 6
  C/C | 2

17. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Stable Disease)
Description: This outcome looks at what genotypes of the GSTP1 c.313A>G (rs1695) gene had stable disease.
Time Frame: 4 years
Population: 11 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 11
participants
  A/A | 8
  A/G | 2
  G/G | 1

18. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Stable Disease)
Description: This outcome looks at what genotypes of the XRCC1 c.1196G>A (rs25487) gene had stable disease.
Time Frame: 4 years
Population: 11 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 11
participants
  A/A | 6
  G/A | 5
  G/G | 0

19. Secondary Outcome: Genetic Polymorphisms That May Alter Treatment Outcomes (Stable Disease)
Description: This outcome looks at what genotypes of the MDR1 c.3435C>T (rs1045642) gene had stable disease.
Time Frame: 4 years
Population: 11 out of 25 participants had a partial response.
Measure: Number; unit: participants
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Number analyzed (Participants) | 11
participants
  C/C | 1
  C/T | 6
  T/T | 4

ADVERSE EVENTS:
Arm/Group | Oxaliplatin/Leucovorin/5-FU
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 20/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin/Leucovorin/5-FU (N=25)
Leukopenia (total WBC) (Investigations) | 13
Neutropenia (Investigations) | 13
Lymphopenia (Investigations) | 8
Anemia (Blood and lymphatic system disorders) | 20
Thrombocytopenia (Investigations) | 12
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 8
Mucositis/stomatitis (Gastrointestinal disorders) | 4
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 8
Blurred vision (Eye disorders) | 3
Allergic reaction/hypersensitivity (Immune system disorders) | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2
AST, SGOT (Investigations) | 11
ALT, SGPT (Investigations) | 12
Sensory neuropathy (Nervous system disorders) | 11
Fatigue (General disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No